CLINICAL TRIAL: NCT03818243
Title: Circadian Character of Food Compulsions and Impulses Control Disorders in Parkinsonian Patients With and Without Resting Leg Syndrome
Acronym: RLS nighfood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHU-421; 2018-A02417-48 (Other: 2018-A02417-48)
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease; Restless Leg Syndrome
Keywords: Parkinson disease; Restless Leg Syndrome; Impulse control disorders; circadian rhythm
MeSH Terms: conditions — Parkinson Disease; Restless Legs Syndrome; Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Intervention Model Description: the 2 groups (patients with Parkinson disease with and without RLS) received the same intervention
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RLS- (Experimental): patients with Parkinson disease without RLS
  Interventions: Behavioral: Diary (for reporting all impulse control disorders especially compulsive eating disorders)
- RLS+ (Experimental): patients with Parkinson disease with RLS
  Interventions: Behavioral: Diary (for reporting all impulse control disorders especially compulsive eating disorders)

INTERVENTIONS:
Behavioral: Diary (for reporting all impulse control disorders especially compulsive eating disorders) — During 7 days, at home, patients must report in their diary all their impulse control disorders especially their compulsive eating disorders. They will detailed each food intake and drink intake and the time.

SUMMARY:
Investigator have recently shown that Parkinson disease patients' with restless leg Syndrome have more frequent impulse control behavior in particular compulsive feeding that patients without Restless Leg Syndrome (RLS).

Investigator hypothesized that presence of RLS in parkinsonian patients could be a risk factor for the emergence of TCI or associated behaviors, occurring preferentially at night.

The main objective of this study is to evaluate in patients with idiopathic Parkinson's disease (IPD) the effect of the presence of a RLS on the evening compulsive eating behavior by studying the circadian modulation of food intake of patients with RLS and impulse control disorders.

For this investigator conduct a prospective study, with 2 groups of Parkinson disease patients (with and without restless leg syndrome), to which investigator have to fill an agenda to know the schedule of the behaviors during the day and the night.

DETAILED DESCRIPTION:
Type of study: prospective, case control study Number of center: 1 (Clermont Ferrand)

Patients:

The study will be performed in 60 patients with Parkinson disease (30 with RLS and 30 without RLS)

Study Performance:

During the first visit (baseline, inclusion visit, 1 hour), each patient will perform an interview about medical history and a neurological examination in order to identify RLS (evaluation using the IRLSSG rating scale).

* Parkinson disease severity will be assessed with the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS UPDRS) and the Hoehn and Yahr scale.
* Cognitive assessment will be evaluated with the Montreal Cognitive assessment (MoCA)
* Blood test to explore plasma ferritin, renal function and plasma glucose. A diary to note all the impulse control behaviour will be given to each patient in order to be completed for the next visit.

Finally, an actimetry system (a watch) will be also provided for each patient in order to record the sleep-wake rhythm and to evaluate the quality and the duration of the sleep.

During the second visit (Baseline + 15 days), each patients will have :

* a neuropsychological assessment (using the Ardouin scale of behavior in Parkinson's disease ASBPD)
* an evaluation of the night eating disorders :
* The night eating syndrome will be evaluated with Night Eating Questionnaire (NEQ)
* The Sleep related eating disorders will be evaluated with the International classification of sleep disorders-third edition criteria
* an evaluation of the Iimpulse control disorder using the questionnaire for impulsive-compulsive disorders in Parkinson's disease rating scale (QUIP RS).
* A sleep and vigilance evaluation using the Epworth scale, the Parkinson's disease sleep scale, the single-question screen for rapid eye movement sleep behavior disorder and the REM sleep behavior disorder screening questionnaire.

Diary and actimetry will be recovered.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 to 80 years
* Patients with a Parkinson disease (PD) with UKPDSBB criteria
* with a medical treatment or other treatment, not modified 4 weeks before inclusion
* Social security affiliation
* Acceptance of the protocol and signature of a written consent

RLS group: Patients with IRLSSG criteria of RLS, with a frequency of RLS ≥ 2 times per week Group without RLS: Patients without IRLSSG criteria of RLS

Exclusion Criteria:

* Patients with an other neurological disease than Parkinson's disease
* Patients with secondary RLS (other than Parkinson's disease)
* Patients with psychiatric diseases
* Patients with cognitive disorder (MoCA <21)
* Patients with body mass index <16.5 or >30
* Patients with sleep-waking rhythm disorders (such as night work…)
* Patients under trusteeship or guardianship or safeguarding of justice

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
The percentage of daily night food intake measured at baseline + 15 day using the diary. | at baseline + 15 day

SECONDARY OUTCOMES:
Percentage of night behavior for the other impulse control disorders , measured at baseline + 15 day using the diary | at baseline + 15 day
Percentage of patients with compulsive food intake measured at baseline + 15 day | at baseline + 15 day
Percentage of patients with others impulse control disorders or other associated behavior measured at baseline + 15 day | at baseline + 15 day
Percentage of patients with the night eating syndrome using the Night Eating Questionnaire measured at baseline + 15 days | at baseline + 15 day
Percentage of patients with Sleep related eating disorders using the International classification of sleep disorders-third edition criteria measured at baseline + 15 days | at baseline + 15 day
sleep caracteristics measured at baseline + 15 days using the accelerometry data | at baseline + 15 day

CONTACTS AND LOCATIONS:
Overall Officials: Ana MARQUES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France